CLINICAL TRIAL: NCT01785979
Title: Prednisone Plus Chloroquine Versus Chloroquine for the Treatment of Hyper-reactive Malarial Splenomegaly in Papua New Guinea: a Randomized Open-label Trial
Brief Title: Prednisone Plus Chloroquine for the Treatment of Hyper-reactive Malarial Splenomegaly
Acronym: LiHMS
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Lihir Medical Centre (Other)
Responsible Party: Principal Investigator, Oriol Mitja, Senior Medical Officer, Lihir Medical Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LiHMS
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Hyper-reactive Malarial Splenomegaly; Malaria; Anaemia
MeSH Terms: conditions — Malaria; Anemia | interventions — Prednisone; Chloroquine; chloroquine diphosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prednisone induction - chloroquine (Experimental): 0.5 mg/Kg daily of prednisone for 4 weeks after randomization, 0.25 mg daily for weeks 5-6, 0.15 mg daily for week 7 and 2.5 mg daily for week 8 and chloroquine at a fixed dose (300 mg base per week) for months 1-12
  Interventions: Drug: prednisone induction - chloroquine
- chloroquine (Active Comparator): chloroquine at a fixed dose (300 mg base per week) for months 1-12
  Interventions: Drug: Chloroquine

INTERVENTIONS:
Drug: prednisone induction - chloroquine — At study entry, the patients will undergo physical examination and laboratory tests, including blood cell count, malaria microscopy, immune-chromatographic test for malaria antigen, malaria serology titers, and serum protein studies with immunoglobulin M quantification, immune-fixation and immunoglobulin free light chains measurement. We will assess all participants at 1, 3, 6 and 12 months after enrollment. Clinical examination and routine laboratory tests are done every 3 months during the follow-up period. Immunoglobulin M quantification and malaria serology are done at baseline, and at month 12 visit.
  Other Names: Deltasone,; Orasone,; Prednicen-M
  Arms: Prednisone induction - chloroquine
Drug: Chloroquine — At study entry, the patients will undergo physical examination and laboratory tests, including blood cell count, malaria microscopy, immune-chromatographic test for malaria antigen, malaria serology titers, and serum protein studies with immunoglobulin M quantification, immune-fixation and immunoglobulin free light chains measurement. We will assess all participants at 1, 3, 6 and 12 months after enrollment. Clinical examination and routine laboratory tests are done every 3 months during the follow-up period. Immunoglobulin M quantification and malaria serology are done at baseline, and at month 12 visit.
  Other Names: Aralen; Resochin; Alchroquin
  Arms: chloroquine

SUMMARY:
This randomized clinical trial will address a complication related to recurrent episodes of malaria in endemic areas - hyper-reactive malarial splenomegaly. We aim to assess the efficacy of chloroquine after prednisone-induction therapy compared to standard treatment of chloroquine alone in the treatment of adult patients with newly diagnosed hyper-reactive malarial splenomegaly.

DETAILED DESCRIPTION:
Hyper-reactive malarious splenomegaly (HMS) is a known chronic autoimmune complication in areas where malaria is endemic. Patients with HMS complain most commonly of abdominal swelling or pain from the enlarged spleen and the condition is defined using clear clinical and laboratory criteria. HMS appears benign in most patients when seen first but if untreated, it leads to severe anaemia and also acute bacterial infections. There is familiar and ethnic clustering suggesting genetic basis. High prevalence rates have been reported in certain areas of Papua New Guinea, and Venezuela, and HMS is also common in parts of sub-Saharan Africa, including Sudan and Ghana.

The treatment of HMS is still empirical since no randomized trials have been done so far. Long term anti-malarial chemoprophylaxis is deemed the mainstay of therapy, but the optimal drug-regimen and duration are unknown. Three to six months may pass before a response is observed, and relapses may occur when therapy is discontinued.

On the basis of the observed benefit in experimental studies, glucocorticoids have been used for severe hyper-reactive malarial splenomegaly in various case reports. Because these cases had a favourable outcome and the drug tolerability was good, prednisone has become an attractive therapeutic option for this disease. Central to the pathophysiology of HMS is the overproduction of Immunoglobulin M due to a functional CD8 T-cell defect and the consequent expansion and activation of B lymphocytes. Glucocorticoids may have an immediate effect due to inhibition of the sequestration of immunoglobulin coated red blood cells by the mononuclear phagocyte system and a later effect due to glucocorticoid-induced inhibition of antibody synthesis. We aim to assess the efficacy of chloroquine after prednisone-induction therapy compared to chloroquine alone in the treatment of adult patients with newly diagnosed hyper-reactive malarial splenomegaly.

ELIGIBILITY:
Inclusion Criteria:

* Defining features of HMS including chronic massive splenomegaly (at least 10 cm below the costal margin); serum Immunoglobulin M elevated more than 3.1 g/L and high malarial antibody titres (above 640).
* Evidence of the polyclonal nature of the lymphocytes by serum immunoglobulin free light chains.
* Aged at least 18 years
* Haemoglobin level of > 5 mg/d

Exclusion Criteria:

* known allergy to chloroquine,
* use of anti-malarial treatment within the preceding month,
* suspected coexisting diseases in which glucocorticoids are contraindicated (e.g. diabetes mellitus, peptic ulcer disease or any acute infection as defined clinically), and
* splenomegaly secondary to known infectious or haematological causes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
composite clinical & immunological endpoint | 12 months
  Clinical cure, defined as a sustained reduction in spleen size of at least 40% at the 12 month follow up examination, compared with the spleen size at the baseline examination. Immunological cure, defined as a two-fold decrease of total immunoglobulin M levels is also needed.

SECONDARY OUTCOMES:
3 months intermediate clinical cure | 3 months
  Reduction in spleen size of at least 40% at the 3 month follow up examination
6 months intermediate clinical cure | 6 months
  Reduction in spleen size of at least 40% at the 3 month follow up examination
Anaemia | 12 months
  Incidence of HMS related-anemia defined by hemoglobin levels below 10 g/L at 12 months
Malaria episode | 12 months
  occurrence of an acute episode of malaria identified by passive-case detection in the hospital facilities during the follow up period.
Bacterial infection | 12 months
  occurrence of an acute bacterial infection identified by passive-case detection in the hospital facilities during the follow up period.

CONTACTS AND LOCATIONS:
Overall Officials: Oriol Mitja, PhD, Principal Investigator — Lihir Medical Centre
Locations (1):
- Lihir medical Centre, Londolovit, New Ireland Province, Papua New Guinea